CLINICAL TRIAL: NCT01032629
Title: A Randomized, Multicenter, Double-Blind, Parallel, Placebo-Controlled Study of the Effects of JNJ-28431754 on Cardiovascular Outcomes in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: CANVAS - CANagliflozin cardioVascular Assessment Study
Acronym: CANVAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016627; 28431754DIA3008 (Other: Janssen Research & Development, LLC); 2009-012140-16 (EudraCT Number)
Record Dates: First submitted 2009-12-10; First posted 2009-12-15 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Risk Factors
Keywords: Diabetes; Type 2 diabetes mellitus; Cardiovascular risk; Cardiovascular outcomes; Canagliflozin (JNJ-28431754); Placebo
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Each patient will receive placebo (inactive medication) on background standard of care for diabetes once daily for the duration of the study
  Interventions: Drug: Placebo
- Canagliflozin (JNJ-28431754) 100 mg (Experimental): Each patient will receive canagliflozin (JNJ-28431754) 100 mg once daily on background standard of care for diabetes once daily for the duration of the study
  Interventions: Drug: Canagliflozin (JNJ-28431754) 100 mg
- Canagliflozin (JNJ-28431754) 300 mg (Experimental): Each patient will receive canagliflozin (JNJ-28431754) 300 mg once daily on background standard of care for diabetes once daily for the duration of the study
  Interventions: Drug: Canagliflozin (JNJ-28431754) 300 mg

INTERVENTIONS:
Drug: Placebo — One placebo capsule taken orally (by mouth) once daily
  Arms: Placebo
Drug: Canagliflozin (JNJ-28431754) 100 mg — One 100 mg capsule taken orally (by mouth) once daily
  Arms: Canagliflozin (JNJ-28431754) 100 mg
Drug: Canagliflozin (JNJ-28431754) 300 mg — One 300 mg capsule taken orally (by mouth) once daily
  Arms: Canagliflozin (JNJ-28431754) 300 mg

SUMMARY:
The study will assess canagliflozin (JNJ-28431754) in the treatment of patients with type 2 diabetes mellitus (T2DM) with regard to cardiovascular (CV) risk for major adverse cardiac events (MACE). Other objectives include evaluating the overall safety, tolerability, and effectiveness of canagliflozin.

The data from this study will be combined with the data from CANVAS-R study (Study of the Effects of Canagliflozin on Renal Endpoints in Adult Subjects with T2DM, NCT01989754) in a pre-specified integrated analysis of CV safety outcomes to satisfy US FDA post-marketing requirements for canagliflozin.

DETAILED DESCRIPTION:
The study will evaluate canagliflozin compared to placebo on CV events including CV death, heart attack, and stroke in patients with T2DM, whose diabetes is not well controlled at the beginning of the study and who have a history of CV events or have a high risk for CV events. The study includes 3 substudies which will compare the effectiveness of lowering blood glucose and assess the safety of canagliflozin relative to placebo in patients receiving specific commonly-used diabetes agents. 4,330 participants will be randomly assigned to treatment with 1 of 2 doses of canagliflozin (100 or 300 mg) or placebo, in a 1:1:1 ratio. This study was originally designed to last for up to 9 years. As per FDA post-marketing requirements for canagliflozin, the study's last subject last visit will now occur when enough MACE events (ie, CV death, nonfatal myocardial infarction, nonfatal stroke) are accumulated between the CANVAS (this study) and CANVAS-R studies. The completion target was reached in February 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes mellitus and greater than or equal to (>=) 30 yrs old with history of cardiovascular (CV) event, or >= 50 yrs old with high risk of CV events
* Patients must have inadequate diabetes control (as defined by glycosylated hemoglobin greater than or equal to 7.0% to less than or equal to 10.5% at screening) and be either (1) not currently on diabetes drug therapy or (2) on therapy with any approved class of diabetes drugs

Exclusion Criteria:

* A history of diabetic ketoacidosis, type 1 diabetes mellitus, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* History of one or more severe hypoglycemic (ie, very low blood sugar) episode within 6 months before screening

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4330 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (305):
- United States (58):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - La Mesa, California
  - Los Gatos, California
  - Pismo Beach, California
  - Stockton, California
  - Walnut Creek, California
  - Doral, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Plantation, Florida
  - Atlanta, Georgia
  - Duluth, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Meridian, Idaho
  - Peoria, Illinois
  - Topeka, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Auburn, Maine
  - Scarborough, Maine
  - Oxon Hill, Maryland
  - Royal Oak, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Camden, New Jersey
  - Flushing, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Gallipolis, Ohio
  - Mentor, Ohio
  - Toledo, Ohio
  - Beaver, Pennsylvania
  - Norristown, Pennsylvania
  - Sayre, Pennsylvania
  - Greenville, South Carolina
  - Kingsport, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Draper, Utah
  - Salt Lake City, Utah
  - Sandy City, Utah
  - West Jordan, Utah
  - Danville, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Argentina (9):
  - Buenos Aires
  - Capital Federal
  - Ciudad Autonma Buenos Aires
  - Corrientes
  - Córdoba
  - Godoy Cruz
  - Mar del Plata
  - Rosario
  - Santa Fe
- Australia (22):
  - Auchenflower
  - Box Hill
  - Caboolture
  - Caringbah
  - Clayton
  - Daw Park
  - East Ringwood
  - Elizabeth Vale
  - Hornsby, Nsw 2077
  - Kippa-Ring
  - Launceston
  - Liverpool
  - Melbourne
  - Milton
  - Parkville
  - Reservoir
  - Sherwood
  - Southport
  - St Leonards
  - West Heidelberg
  - Wollongong
  - Woolloongabba
- Belgium (6):
  - Arlon
  - Bonheiden
  - Brussels
  - Edegem
  - Genk
  - Leuven
- Canada (16):
  - Calgary, Alberta
  - Coquitlam, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Nemarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Lévis, Quebec
  - Montreal, Quebec
  - Val-Bélair, Quebec
  - Saskatoon, Saskatchewan
- Colombia (2):
  - Bogotá
  - Floridablanca
- Czechia (7):
  - Kralupy nad Vltavou
  - Moravský Krumlov
  - Olomouc
  - Ostrava
  - Písek
  - Prague
  - Znojmo
- Estonia (4):
  - Pärnu
  - Tallinn
  - Tartu
  - Viljandi
- France (3):
  - Amiens
  - Nîmes
  - Pessac
- Germany (11):
  - Berlin
  - Dortmund
  - Dresden
  - Hamburg
  - Künzing
  - Mainz
  - Münster
  - Pirna
  - Saarlouis
  - Speyer
  - Villingen-Schwenningen
- Hungary (4):
  - Budapest
  - Kecskemét
  - Mosonmagyaróvár
  - Zalaegerszeg
- India (31):
  - Ahemadabad
  - Ahmedabad
  - Ambawadi
  - Bangalore
  - Bangalore, Karnataka
  - Belagavi
  - Calicut
  - Chennai
  - Coimbatore
  - Ernākulam
  - Ghaziabad
  - Hyderabad
  - Indore
  - Jaipur
  - Karnāl
  - Kerala
  - Kochi
  - Kolkata
  - Lucknow
  - Mangalore
  - Mumbai
  - Mysore
  - Nagpur
  - New Delhi
  - Patna
  - Pune
  - Rajkot
  - Trivandrum, Kerala
  - Vadodhara
  - Vijayawada
  - Visakhapatnam
- Israel (4):
  - Beersheba
  - Holon
  - Jerusalem
  - Kfar Saba
- Luxembourg, Luxembourg
- Malaysia (7):
  - George Town
  - Johor Bahru
  - Kota Bharu
  - Kuala Lumpur
  - Petaling Jaya
  - Pulau Pinang
  - Subang Jaya
- Mexico (6):
  - Aguascalientes
  - Celaya
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey
- Netherlands (16):
  - Almelo
  - Almere Stad
  - Amsterdam
  - Arnhem
  - Delft
  - Den Helder
  - Dordrecht
  - Eindhoven
  - Groningen
  - Hoorn
  - Rotterdam
  - Tilburg
  - Utrecht
  - Velp Gld
  - Zoetermeer
  - Zwijndrecht
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Tauranga
  - Wellington
- Norway (9):
  - Asker
  - Ålesund
  - Bekkestua
  - Elverum
  - Hamar
  - Lierskogen
  - Moss
  - Oslo
  - Skedsmokorset
- Poland (14):
  - Bialystok
  - Ciechocinek
  - Gniewkowo
  - Grudziądz
  - Katowice
  - Krakow
  - Lublin
  - Poznan
  - Płock
  - Rzeszów
  - Sławków
  - Torun
  - Warsaw
  - Wroclaw
- Russia (22):
  - Arkhangelsk
  - Chelyabinsk
  - Kemerovo
  - Kirov
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Penza
  - Rostov-on-Don
  - Russia
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tomsk
  - Tula
  - Tyumen
  - Yaroslavl
  - Yaroslavl Nap
  - Yekaterinburg
- Spain (14):
  - Alicante
  - Almería
  - Barcelona
  - Figueres
  - Madrid
  - Málaga
  - Oviedo
  - Reus
  - Sabadell
  - Sant Joan d'Alacant
  - Santiago de Compostela
  - Seville
  - Valencia
  - Viladecans
- Sweden (9):
  - Borås
  - Gothenburg
  - Helsingborg
  - Lund
  - Malmo
  - Oskarshamn
  - Piteå
  - Stockholm
  - Uddevalla
- Ukraine (10):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Odesa
  - Ternopil
  - Uzhhorod
  - Vinnitsa
  - Zaporizhzhya
- United Kingdom (15):
  - Belfast
  - Blackburn
  - Bolton
  - Chorley
  - Derby
  - Glasgow
  - Hull
  - Leicester
  - Liverpool
  - London
  - Londonderry
  - Manchester
  - Randalstown
  - Salford
  - York

REFERENCES:
- [Derived] Mottl A, Scott C, Green JB, Heerspink HJL, Mann JFE, McGill JB, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Vaduganathan M, Agarwal R; CONFIDENCE Trial Investigators. Baseline Kidney Function, Albuminuria, and Urine Albumin-Creatinine Ratio Reduction with Finerenone, Empagliflozin, or Both: Post Hoc Analyses of CONFIDENCE Trial. J Am Soc Nephrol. 2025 Nov 6. doi: 10.1681/ASN.0000000928. Online ahead of print. No abstract available. PMID 41196655
- [Derived] Bayes-Genis A, Cai A, Liu Y, Pandey A, Pop-Busui R, Hansen M, Januzzi JL. Impact of canagliflozin on heart stress and outcomes: Pooled insights from CREDENCE and CANVAS. Eur J Heart Fail. 2025 Dec;27(12):2887-2896. doi: 10.1002/ejhf.3786. Epub 2025 Jul 21. PMID 40689549
- [Derived] Doi Y, Hamano T, Yamaguchi O, Isaka Y. Canagliflozin may increase thromboembolic events in males with erythrocytosis but not in females. Blood Adv. 2025 Jul 8;9(13):3202-3212. doi: 10.1182/bloodadvances.2025016320. PMID 40239057
- [Derived] Nguyen TN, Yu J, Perkovic V, Jardine M, Mahaffey KW, Chow CK, Arnott C, Lindley RI. The Efficacy and Safety of Canagliflozin by Frailty Status in Participants of the CANVAS and CREDENCE Trials. J Am Geriatr Soc. 2025 Jun;73(6):1787-1796. doi: 10.1111/jgs.19444. Epub 2025 Mar 19. PMID 40105285
- [Derived] Chatur S, Vaduganathan M, Fletcher RA, Perkovic V, Heerspink H, Arnott C, Pollock C, Mahaffey KW, Neal B, Jardine M, Solomon SD, Neuen BL. Canagliflozin reduces oral loop diuretic intensification in patients with type 2 diabetes: A participant-level pooled analysis of the CANVAS and CREDENCE trials. Eur J Heart Fail. 2025 Jun;27(6):994-1002. doi: 10.1002/ejhf.3586. Epub 2025 Jan 23. PMID 39844714
- [Derived] Vaduganathan M, Cannon CP, Jardine MJ, Heerspink HJL, Arnott C, Neuen BL, Sarraju A, Gogate J, Seufert J, Neal B, Perkovic V, Mahaffey KW, Kosiborod MN. Effects of canagliflozin on total heart failure events across the kidney function spectrum: Participant-level pooled analysis from the CANVAS Program and CREDENCE trial. Eur J Heart Fail. 2024 Sep;26(9):1967-1975. doi: 10.1002/ejhf.3292. Epub 2024 Jun 26. PMID 38932575
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Sharma A, Razaghizad A, Joury A, Levin A, Bajaj HS, Mancini GBJ, Wong NC, Slee A, Ang FG, Rapattoni W, Neuen BL, Arnott C, Perkovic V, Mahaffey KW. Primary and Secondary Cardiovascular and Kidney Prevention With Canagliflozin: Insights From the CANVAS Program and CREDENCE Trial. J Am Heart Assoc. 2024 Feb 6;13(3):e031586. doi: 10.1161/JAHA.123.031586. Epub 2024 Jan 19. PMID 38240199
- [Derived] Yu J, Sweeting AN, Gianacas C, Houston L, Lee V, Fletcher RA, Perkovic V, Li Q, Neuen BL, Berwanger O, Heerspink HJL, de Zeeuw D, Arnott C. The effects of canagliflozin in type 2 diabetes in subgroups defined by population-specific body mass index: Insights from the CANVAS Program and CREDENCE trial. Diabetes Obes Metab. 2023 Dec;25(12):3724-3735. doi: 10.1111/dom.15267. Epub 2023 Sep 6. PMID 37671609
- [Derived] Sen T, Ju W, Nair V, Ladd P, Menon R, Otto EA, Pyle L, Vigers T, Nelson RG, Arnott C, Neal B, Hansen MK, Kretzler M, Bjornstad P, Heerspink HJL. Sodium glucose co-transporter 2 inhibition increases epidermal growth factor expression and improves outcomes in patients with type 2 diabetes. Kidney Int. 2023 Oct;104(4):828-839. doi: 10.1016/j.kint.2023.07.007. Epub 2023 Aug 4. PMID 37543256
- [Derived] Fletcher RA, Arnott C, Rockenschaub P, Schutte AE, Carpenter L, Vaduganathan M, Agarwal R, Bakris G, Chang TI, Heerspink HJL, Jardine MJ, Mahaffey KW, Neal B, Pollock C, Jun M, Rodgers A, Perkovic V, Neuen BL. Canagliflozin, Blood Pressure Variability, and Risk of Cardiovascular, Kidney, and Mortality Outcomes: Pooled Individual Participant Data From the CANVAS and CREDENCE Trials. J Am Heart Assoc. 2023 Jul 4;12(13):e028516. doi: 10.1161/JAHA.122.028516. Epub 2023 Jun 22. PMID 37345834
- [Derived] Borisov AN, Kutz A, Christ ER, Heim MH, Ebrahimi F. Canagliflozin and Metabolic Associated Fatty Liver Disease in Patients With Diabetes Mellitus: New Insights From CANVAS. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2940-2949. doi: 10.1210/clinem/dgad249. PMID 37149821
- [Derived] Ferrannini G, Pollock C, Natali A, Yavin Y, Mahaffey KW, Ferrannini E. Extremes of both weight gain and weight loss are associated with increased incidence of heart failure and cardiovascular death: evidence from the CANVAS Program and CREDENCE. Cardiovasc Diabetol. 2023 Apr 29;22(1):100. doi: 10.1186/s12933-023-01832-5. PMID 37120538
- [Derived] Rasmussen DGK, Hansen MK, Blair J, Jatkoe TA, Neal B, Karsdal MA, Genovese F. Endotrophin is a risk marker of complications in CANagliflozin cardioVascular Assessment Study (CANVAS): a randomized controlled trial. Cardiovasc Diabetol. 2022 Nov 28;21(1):261. doi: 10.1186/s12933-022-01666-7. PMID 36443792
- [Derived] Nunes JC, Yu J, Arnott C, Jardine MJ, Perkovic V, Mahaffey KW. Canagliflozin, mental health adverse events and diabetes: Exploratory analysis of the CREDENCE trial and CANVAS Program. Diabetes Obes Metab. 2022 Dec;24(12):2459-2464. doi: 10.1111/dom.14832. Epub 2022 Aug 19. No abstract available. PMID 35938182
- [Derived] Ferrannini E, Baldi S, Scozzaro T, Tsimihodimos V, Tesfaye F, Shaw W, Rosenthal N, Figtree GA, Neal B, Mahaffey KW, Perkovic V, Hansen MK. Fasting Substrate Concentrations Predict Cardiovascular Outcomes in the CANagliflozin cardioVascular Assessment Study (CANVAS). Diabetes Care. 2022 Aug 1;45(8):1893-1899. doi: 10.2337/dc21-2398. PMID 35724306
- [Derived] Vaduganathan M, Sattar N, Xu J, Butler J, Mahaffey KW, Neal B, Shaw W, Rosenthal N, Pfeifer M, Hansen MK, Januzzi JL Jr. Stress Cardiac Biomarkers, Cardiovascular and Renal Outcomes, and Response to Canagliflozin. J Am Coll Cardiol. 2022 Feb 8;79(5):432-444. doi: 10.1016/j.jacc.2021.11.027. PMID 35115099
- [Derived] Waijer SW, Sen T, Arnott C, Neal B, Kosterink JGW, Mahaffey KW, Parikh CR, de Zeeuw D, Perkovic V, Neuen BL, Coca SG, Hansen MK, Gansevoort RT, Heerspink HJL. Association between TNF Receptors and KIM-1 with Kidney Outcomes in Early-Stage Diabetic Kidney Disease. Clin J Am Soc Nephrol. 2022 Feb;17(2):251-259. doi: 10.2215/CJN.08780621. Epub 2021 Dec 7. PMID 34876454
- [Derived] Young TK, Li JW, Kang A, Heerspink HJL, Hockham C, Arnott C, Neuen BL, Zoungas S, Mahaffey KW, Perkovic V, de Zeeuw D, Fulcher G, Neal B, Jardine M. Effects of canagliflozin compared with placebo on major adverse cardiovascular and kidney events in patient groups with different baseline levels of HbA1c, disease duration and treatment intensity: results from the CANVAS Program. Diabetologia. 2021 Nov;64(11):2402-2414. doi: 10.1007/s00125-021-05524-1. Epub 2021 Aug 26. PMID 34448033
- [Derived] Yu J, Li J, Leaver PJ, Arnott C, Huffman MD, Udell JA, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Rosenthal N, Neal B, Figtree GA. Effects of canagliflozin on myocardial infarction: a post hoc analysis of the CANVAS programme and CREDENCE trial. Cardiovasc Res. 2022 Mar 16;118(4):1103-1114. doi: 10.1093/cvr/cvab128. PMID 33826709
- [Derived] Yu J, Arnott C, Neuen BL, Heersprink HL, Mahaffey KW, Cannon CP, Khan SS, Baldridge AS, Shah SJ, Huang Y, Li C, Figtree GA, Perkovic V, Jardine MJ, Neal B, Huffman MD. Cardiovascular and renal outcomes with canagliflozin according to baseline diuretic use: a post hoc analysis from the CANVAS Program. ESC Heart Fail. 2021 Apr;8(2):1482-1493. doi: 10.1002/ehf2.13236. Epub 2021 Feb 17. PMID 33595905
- [Derived] Januzzi JL Jr, Butler J, Sattar N, Xu J, Shaw W, Rosenthal N, Pfeifer M, Mahaffey KW, Neal B, Hansen MK. Insulin-Like Growth Factor Binding Protein 7 Predicts Renal and Cardiovascular Outcomes in the Canagliflozin Cardiovascular Assessment Study. Diabetes Care. 2021 Jan;44(1):210-216. doi: 10.2337/dc20-1889. Epub 2020 Nov 6. PMID 33158949
- [Derived] Januzzi JL Jr, Xu J, Li J, Shaw W, Oh R, Pfeifer M, Butler J, Sattar N, Mahaffey KW, Neal B, Hansen MK. Effects of Canagliflozin on Amino-Terminal Pro-B-Type Natriuretic Peptide: Implications for Cardiovascular Risk Reduction. J Am Coll Cardiol. 2020 Nov 3;76(18):2076-2085. doi: 10.1016/j.jacc.2020.09.004. PMID 33121714
- [Derived] Neuen BL, Ohkuma T, Neal B, Matthews DR, de Zeeuw D, Mahaffey KW, Fulcher G, Blais J, Li Q, Jardine MJ, Perkovic V, Wheeler DC. Relative and Absolute Risk Reductions in Cardiovascular and Kidney Outcomes With Canagliflozin Across KDIGO Risk Categories: Findings From the CANVAS Program. Am J Kidney Dis. 2021 Jan;77(1):23-34.e1. doi: 10.1053/j.ajkd.2020.06.018. Epub 2020 Sep 21. PMID 32971190
- [Derived] Oshima M, Neal B, Toyama T, Ohkuma T, Li Q, de Zeeuw D, Heerspink HJL, Mahaffey KW, Fulcher G, Canovatchel W, Matthews DR, Perkovic V. Different eGFR Decline Thresholds and Renal Effects of Canagliflozin: Data from the CANVAS Program. J Am Soc Nephrol. 2020 Oct;31(10):2446-2456. doi: 10.1681/ASN.2019121312. Epub 2020 Jul 21. PMID 32694216
- [Derived] Matthews DR, Wysham C, Davies M, Slee A, Alba M, Lee M, Perkovic V, Mahaffey KW, Neal B. Effects of canagliflozin on initiation of insulin and other antihyperglycaemic agents in the CANVAS Program. Diabetes Obes Metab. 2020 Nov;22(11):2199-2203. doi: 10.1111/dom.14143. Epub 2020 Aug 24. PMID 32691499
- [Derived] Zhou Z, Jardine M, Perkovic V, Matthews DR, Mahaffey KW, de Zeeuw D, Fulcher G, Desai M, Oh R, Simpson R, Watts NB, Neal B. Canagliflozin and fracture risk in individuals with type 2 diabetes: results from the CANVAS Program. Diabetologia. 2019 Oct;62(10):1854-1867. doi: 10.1007/s00125-019-4955-5. Epub 2019 Aug 10. PMID 31399845
- [Derived] Figtree GA, Radholm K, Barrett TD, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Neal B. Effects of Canagliflozin on Heart Failure Outcomes Associated With Preserved and Reduced Ejection Fraction in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2591-2593. doi: 10.1161/CIRCULATIONAHA.119.040057. Epub 2019 Mar 17. No abstract available. PMID 30882240
- [Derived] Zhou Z, Lindley RI, Radholm K, Jenkins B, Watson J, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Shaw W, Oh R, Desai M, Matthews DR, Neal B. Canagliflozin and Stroke in Type 2 Diabetes Mellitus. Stroke. 2019 Feb;50(2):396-404. doi: 10.1161/STROKEAHA.118.023009. PMID 30591006
- [Derived] Neuen BL, Ohkuma T, Neal B, Matthews DR, de Zeeuw D, Mahaffey KW, Fulcher G, Desai M, Li Q, Deng H, Rosenthal N, Jardine MJ, Bakris G, Perkovic V. Cardiovascular and Renal Outcomes With Canagliflozin According to Baseline Kidney Function. Circulation. 2018 Oct 9;138(15):1537-1550. doi: 10.1161/CIRCULATIONAHA.118.035901. PMID 29941478
- [Derived] Perkovic V, de Zeeuw D, Mahaffey KW, Fulcher G, Erondu N, Shaw W, Barrett TD, Weidner-Wells M, Deng H, Matthews DR, Neal B. Canagliflozin and renal outcomes in type 2 diabetes: results from the CANVAS Program randomised clinical trials. Lancet Diabetes Endocrinol. 2018 Sep;6(9):691-704. doi: 10.1016/S2213-8587(18)30141-4. Epub 2018 Jun 21. PMID 29937267
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Eligibility varies among the 4 sodium-glucose cotransporter-2 inhibitor cardiovascular outcomes trials: implications for the general type 2 diabetes US population. Am J Manag Care. 2018 Apr;24(8 Suppl):S138-S145. PMID 29693360
- [Derived] Radholm K, Figtree G, Perkovic V, Solomon SD, Mahaffey KW, de Zeeuw D, Fulcher G, Barrett TD, Shaw W, Desai M, Matthews DR, Neal B. Canagliflozin and Heart Failure in Type 2 Diabetes Mellitus: Results From the CANVAS Program. Circulation. 2018 Jul 31;138(5):458-468. doi: 10.1161/CIRCULATIONAHA.118.034222. PMID 29526832
- [Derived] Mahaffey KW, Neal B, Perkovic V, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Fabbrini E, Sun T, Li Q, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin for Primary and Secondary Prevention of Cardiovascular Events: Results From the CANVAS Program (Canagliflozin Cardiovascular Assessment Study). Circulation. 2018 Jan 23;137(4):323-334. doi: 10.1161/CIRCULATIONAHA.117.032038. Epub 2017 Nov 13. PMID 29133604
- [Derived] Yale JF, Xie J, Sherman SE, Garceau C. Canagliflozin in Conjunction With Sulfonylurea Maintains Glycemic Control and Weight Loss Over 52 Weeks: A Randomized, Controlled Trial in Patients With Type 2 Diabetes Mellitus. Clin Ther. 2017 Nov;39(11):2230-2242.e2. doi: 10.1016/j.clinthera.2017.10.003. Epub 2017 Nov 3. PMID 29103664
- [Derived] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Gavin JR 3rd, Davies MJ, Davies M, Vijapurkar U, Alba M, Meininger G. The efficacy and safety of canagliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015;31(9):1693-702. doi: 10.1185/03007995.2015.1067192. Epub 2015 Sep 4. PMID 26121561
- [Derived] Fulcher G, Matthews DR, Perkovic V, de Zeeuw D, Mahaffey KW, Weiss R, Rosenstock J, Capuano G, Desai M, Shaw W, Vercruysse F, Meininger G, Neal B. Efficacy and Safety of Canagliflozin Used in Conjunction with Sulfonylurea in Patients with Type 2 Diabetes Mellitus: A Randomized, Controlled Trial. Diabetes Ther. 2015 Sep;6(3):289-302. doi: 10.1007/s13300-015-0117-z. Epub 2015 Jun 17. PMID 26081793
- [Derived] Neal B, Perkovic V, de Zeeuw D, Mahaffey KW, Fulcher G, Ways K, Desai M, Shaw W, Capuano G, Alba M, Jiang J, Vercruysse F, Meininger G, Matthews D; CANVAS Trial Collaborative Group. Efficacy and safety of canagliflozin, an inhibitor of sodium-glucose cotransporter 2, when used in conjunction with insulin therapy in patients with type 2 diabetes. Diabetes Care. 2015 Mar;38(3):403-11. doi: 10.2337/dc14-1237. Epub 2014 Dec 2. PMID 25468945
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339
- [Derived] Neal B, Perkovic V, de Zeeuw D, Mahaffey KW, Fulcher G, Stein P, Desai M, Shaw W, Jiang J, Vercruysse F, Meininger G, Matthews D. Rationale, design, and baseline characteristics of the Canagliflozin Cardiovascular Assessment Study (CANVAS)--a randomized placebo-controlled trial. Am Heart J. 2013 Aug;166(2):217-223.e11. doi: 10.1016/j.ahj.2013.05.007. Epub 2013 Jun 24. PMID 23895803

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No Text enterred
Groups:
- Placebo: Participants received one placebo capsule orally once daily for the duration of the study or until early discontinuation from treatment.
- Canagliflozin 100 mg: Participants received one canagliflozin 100 milligram (mg) capsule once daily for the duration of the study or until early discontinuation from treatment.
- Canagliflozin 300 mg: Participants received one canagliflozin 300 mg capsule once daily for the duration of the study or until early discontinuation from treatment.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 1442 | 1445 | 1443
Treated | 1441 | 1445 | 1441
Completed | 1297 (Participants who died on trial were considered completed) | 1344 (Participants who died on trial were considered completed) | 1355 (Participants who died on trial were considered completed)
Not Completed | 145 | 101 | 88
Not completed — Closed Site | 21 | 18 | 16
Not completed — Withdrawal by Subject | 50 | 36 | 35
Not completed — Lost to Follow-up | 74 | 47 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 1442 | 1445 | 1443 | 4330
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (7.94) | 62.2 (8) | 62.8 (8.13) | 62.4 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486 | 484 | 499 | 1469
  Male | 956 | 961 | 944 | 2861
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 149 | 142 | 125 | 416
  Not Hispanic or Latino | 1288 | 1300 | 1317 | 3905
  Unknown or Not Reported | 5 | 3 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 1 | 5
  Asian | 262 | 270 | 263 | 795
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3 | 6
  Black or African American | 35 | 32 | 38 | 105
  White | 1064 | 1060 | 1055 | 3179
  More than one race | 10 | 8 | 13 | 31
  Unknown or Not Reported | 67 | 72 | 70 | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 262 | 270 | 263 | 795
  Black or African American | 35 | 32 | 38 | 105
  Hispanic or Latino | 134 | 123 | 106 | 363
  Other | 82 | 86 | 88 | 256
  White Non- Hispanic | 929 | 934 | 948 | 2811
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 57 | 48 | 55 | 160
  Australia | 57 | 60 | 60 | 177
  Belgium | 3 | 10 | 8 | 21
  Canada | 134 | 139 | 123 | 396
  Colombia | 4 | 1 | 2 | 7
  Czech Republic | 37 | 37 | 43 | 117
  Estonia | 19 | 13 | 12 | 44
  Germany | 47 | 62 | 66 | 175
  Hungary | 38 | 50 | 37 | 125
  India | 229 | 232 | 234 | 695
  Israel | 5 | 11 | 9 | 25
  Luxembourg | 1 | 0 | 0 | 1
  Malaysia | 32 | 24 | 17 | 73
  Mexico | 40 | 48 | 36 | 124
  Netherlands | 70 | 77 | 81 | 228
  New Zealand | 27 | 22 | 25 | 74
  Norway | 41 | 33 | 35 | 109
  Poland | 47 | 54 | 43 | 144
  Russia | 146 | 118 | 125 | 389
  Spain | 64 | 74 | 71 | 209
  Sweden | 23 | 26 | 22 | 71
  Ukraine | 50 | 39 | 58 | 147
  United Kingdom | 31 | 29 | 32 | 92
  United States | 240 | 238 | 249 | 727

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiovascular Events (MACE) Composite of Cardiovascular (CV) Death, Non-Fatal Myocardial Infarction (MI), and Non-Fatal Stroke
Description: MACE, defined as a composite of CV death, non-fatal MI, and nonfatal stroke. Adjudication of these events by the Endpoint Adjudication Committee (EAC) was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of MACE are presented.
Time Frame: Up to approximately 8 years
Population: The primary analysis was based on the intent-to-treat (ITT) analysis set for adjudicated MACE, and included all randomized participants. As per planned analysis, the results were reported separately and combined for both doses.
Measure: Number; unit: Events per 1000 patient-year
Groups:
- Canagliflozin (Total): Participants received one canagliflozin 100 mg or 300 mg capsule once daily for the duration of the study or until early discontinuation from treatment.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Canagliflozin (Total)
Number analyzed (Participants) | 1442 | 1445 | 1443 | 2888
Events per 1000 patient-year | 30.36 | 28.41 | 25.37 | 26.89
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.4576, Cox proportional hazard model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.78 to 1.12]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0467, Cox proportional hazard model; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.00]
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin (Total); Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.1120, Cox proportional hazard method; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.75 to 1.03]

2. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Steady-State Beta-Cell Function (HOMA2-%B) at the End-of-Treatment (EOT)
Description: The homeostatic model assessment (HOMA) quantifies insulin resistance and beta-cell function. HOMA2-%B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady-state beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100 percent.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) included subset of participants who were not receiving insulin at baseline and had at least one post-baseline HOMA2-%B measurement on-treatment prior to initiation of insulin.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HOMA2
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 463 | 511 | 477
Percentage of HOMA2 | 4.02 (1.611) | 6.82 (1.533) | 8.09 (1.587)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.210, ANCOVA; Difference of Least Square Mean = 2.79, 95% CI 2-sided [-1.571 to 7.154], Standard Error of Mean 2.224
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.072, ANCOVA; Difference of Least Square Mean = 4.07, 95% CI 2-sided [-0.368 to 8.504], Standard Error of Mean 2.261

3. Secondary Outcome: Percentage of Participants With Progression of Albuminuria at the End-of-Treatment
Description: Progression defined as the development of micro-albuminuria (albumin/creatinine ratio (ACR) greater than or equal to [>=] 30 milligram per gram (mg/g) and less than or equal to <= 300 mg/g) or macroalbuminuria (ACR of >300 mg/g) in a participant with baseline normoalbuminuria or the development of macro-albuminuria in a participant with baseline microalbuminuria. Percentage of participants with progression of albuminuria at the end-of-treatment were assessed.
Time Frame: End of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were treated, had both baseline and post-baseline ACR measurements, and baseline ACR<=300 mg/g.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1286 | 1334 | 1298
Percentage of participants | 24.0 | 20.2 | 18.3
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.67 to 0.97]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.58 to 0.85]

4. Secondary Outcome: Change From Baseline in Proinsulin/Insulin (PI/I) Ratio at the End-of-Treatment
Description: A raised proinsulin-to-insulin ratio due to impaired processing of proinsulin is an early marker of beta cell dysfunction. Beta-cell dysfunction was evaluated by calculating the PI/I ratio, which estimates the capacity of beta cells to convert proinsulin to insulin and may represent an acceptable method to indicate the degree of beta-cell secretion.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set: all randomized participants who received at least 1 dose of study drug. 'N' (number of participants analyzed): number of participants evaluable for this outcome measure, had both baseline and any post-baseline PI/I ratio measurements on-treatment prior to initiation of insulin and didn't receive insulin through baseline.
Measure: Least Squares Mean (Standard Error); unit: Picomole per milli international units
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 370 | 426 | 412
Picomole per milli international units | 0.70 (0.150) | 0.67 (0.140) | 1.03 (0.142)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.03, 95% CI 2-sided [-0.429 to 0.374], Standard Error of Mean 0.205
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.33, 95% CI 2-sided [-0.079 to 0.731], Standard Error of Mean 0.206

5. Secondary Outcome: Change From Baseline in Urinary Albumin/Creatinine Ratio at End-of-Treatment
Description: Urinary Albumin/Creatinine Ratio is a potential marker of chronic kidney disease, calculated as a ratio of Urinary Albumin and Urinary Creatinine.
Time Frame: Baseline and End of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and had both baseline and post-baseline ACR measurements.
Measure: Geometric Mean (95% Confidence Interval); unit: Milligram per gram (mg/g)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1377 | 1398 | 1384
Milligram per gram (mg/g) | 29.30 [27.66 to 31.03] | 25.50 [24.09 to 27] | 24.47 [23.11 to 25.91]
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Geometric mean ratio = 0.87, 95% CI 2-sided [0.800 to 0.940]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Geometric mean ratio = 0.84, 95% CI 2-sided [0.770 to 0.910]

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at End-of-Treatment
Description: Change from baseline in Estimated Glomerular Filtration Rate (eGFR) was assessed at end of treatment. GFR is a measure of the rate at which blood is filtered by the kidney. Modification of Diet in Renal Disease (MDRD) is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and sex. eGFR milliliters/minute/1.73 meters square (mL/min/1.73 m^2) = 175 * (serum creatinine) ^ 1.154 * (Age) ^-0.203 *(0.742 if female) * (1.21 if Black).
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure who had both baseline and post-baseline eGFR measurements.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1394 | 1412 | 1383
mL/min/1.73 m^2 | -5.23 (0.390) | -3.55 (0.388) | -3.98 (0.392)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 1.68, 95% CI 2-sided [0.599 to 2.755], Standard Error of Mean 0.550
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 1.24, 95% CI 2-sided [0.160 to 2.328], Standard Error of Mean 0.553

7. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at End-of-Treatment
Description: Change from baseline in glycated hemoglobin (HbA1c) percentage (%) was assessed at end of treatment. Glycated hemoglobin is a form of hemoglobin that is measured primarily to identify the average glucose concentration in the blood.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure who had both baseline and any post-baseline HbA1C measurements.
Measure: Least Squares Mean (Standard Error); unit: HbA1c (%)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1366 | 1392 | 1352
HbA1c (%) | 0.01 (0.032) | -0.26 (0.032) | -0.31 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.27, 95% CI 2-sided [-0.355 to -0.177], Standard Error of Mean 0.045
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.32, 95% CI 2-sided [-0.405 to -0.227], Standard Error of Mean 0.046

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Levels at End-of-Treatment
Description: Change from baseline in the fasting plasma glucose levels at end-of-treatment was assessed.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and had both baseline and post-baseline fasting plasma glucose measurements.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1392 | 1410 | 1377
Millimoles per liter (mmol/L) | 0.16 (0.076) | -0.42 (0.075) | -0.57 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.58, 95% CI 2-sided [-0.794 to -0.374], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.73, 95% CI 2-sided [-0.945 to -0.523], Standard Error of Mean 0.108

9. Secondary Outcome: Percent Change From Baseline in Body Weight at End-of-Treatment
Description: Percent change from baseline in body weight was assessed at the end of treatment.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and who had both baseline and post-baseline body weight.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1398 | 1415 | 1388
Percent change | -0.50 (0.184) | -3.47 (0.183) | -4.12 (0.185)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -2.96, 95% CI [-3.472 to -2.454], Standard Error of Mean 0.260
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -3.61, 95% CI 2-sided [-4.125 to -3.103], Standard Error of Mean 0.261

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at End-of-Treatment
Description: Change from baseline in systolic blood pressure and diastolic blood pressure was assessed.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure who and had both baseline and post-baseline blood pressure measurements.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1398 | 1415 | 1388
Millimeter of mercury (mmHg)
  SBP(Change at end of treatment) | -1.96 (0.377) | -4.91 (0.375) | -6.49 (0.378)
  DBP (Change at end of treatment) | -2.88 (0.223) | -3.70 (0.221) | -4.51 (0.223)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Statistical analysis (Systolic blood pressure) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -2.96, 95% CI 2-sided [-3.998 to -1.914], Standard Error of Mean 0.532
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Statistical analysis (Systolic blood pressure) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -4.53, 95% CI 2-sided [-5.579 to -3.484], Standard Error of Mean 0.534
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 100 mg; Statistical analysis (Diastolic blood pressure) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -0.82, 95% CI 2-sided [-1.437 to -0.205], Standard Error of Mean 0.314
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg; Statistical analysis (Diastolic blood pressure) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = -1.63, 95% CI 2-sided [-2.245 to -1.007], Standard Error of Mean 0.316

11. Secondary Outcome: Change From Baseline in Triglycerides Levels at End-of-Treatment
Description: Change from baseline in triglycerides levels was assessed.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: On-treatment set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and who had both baseline and post-baseline lipid measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1325 | 1371 | 1321
mmol/L | 0.05 (1.597) | 0.13 (1.679) | 0.09 (1.238)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Hodges-Lehman Estimate = 0.02, 95% CI 2-sided [-0.040 to 0.070]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Other; Hodges-Lehman Estimate = 0.02, 95% CI 2-sided [-0.030 to 0.080]

12. Secondary Outcome: Change From Baseline in Cholesterol, High-Density Lipoprotein Cholesterol (HDL-C) and Low Density Lipoprotein Cholesterol (LDL-C) Levels at End-of-Treatment
Description: Change from baseline in cholesterol, high-density lipoprotein cholesterol and low density lipoprotein cholesterol levels were assessed.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1325 | 1371 | 1321
mmol/L
  Cholesterol (change at EOT) | -0.07 (0.028) | 0.11 (0.027) | 0.16 (0.028)
  HDL-C (change at EOT) | -0.01 (0.006) | 0.04 (0.006) | 0.05 (0.006)
  LDL-C (change at EOT) | -0.07 (0.022) | 0.04 (0.022) | 0.10 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Statistical analysis (Cholesterol) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.18, 95% CI 2-sided [0.105 to 0.259], Standard Error of Mean 0.039
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Statistical analysis (Cholesterol) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.23, 95% CI 2-sided [0.152 to 0.307], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 100 mg; Statistical analysis (HDL-C); Test type: Other; Difference of Least Square Mean = 0.05, 95% CI 2-sided [0.031 to 0.065], Standard Error of Mean 0.009
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg; Statistical analysis (HDL-C) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.06, 95% CI 2-sided [0.040 to 0.075], Standard Error of Mean 0.009
Statistical Analysis 5: Comparison: Placebo vs Canagliflozin 100 mg; Statistical analysis (LDL-C) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.11, 95% CI 2-sided [0.046 to 0.170], Standard Error of Mean 0.032
Statistical Analysis 6: Comparison: Placebo vs Canagliflozin 300 mg; Statistical analysis (LDL-C) Comparison for canagliflozin versus placebo is reported here; Test type: Other; Difference of Least Square Mean = 0.16, 95% CI 2-sided [0.102 to 0.226], Standard Error of Mean 0.032

13. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) to High-Density Lipoprotein-Cholesterol (HDL-C) Ratio at End-of-Treatment
Description: Change from baseline in LDL-C to HDL-C ratio was assessed.
Time Frame: Baseline and end of treatment (approximately 338 weeks)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 1325 | 1371 | 1321
Ratio | -0.04 (0.021) | -0.02 (0.021) | 0.00 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Other; Difference of Least Square Mean = 0.02, 95% CI 2-sided [-0.040 to 0.076], Standard Error of Mean 0.030
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Other; Difference of Least Square Mean = 0.04, 95% CI 2-sided [-0.023 to 0.094], Standard Error of Mean 0.030

ADVERSE EVENTS:
Time Frame: Approximately 8 years
Description: On-treatment analysis set included all randomized participants who were treated and received at least 1 dose of study drug.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
All-Cause Mortality (participants affected / at risk) | 74/1441 | 68/1445 | 66/1441
Serious Adverse Events (participants affected / at risk) | 584/1441 | 601/1445 | 606/1441
Other Adverse Events (participants affected / at risk) | 1137/1441 | 1146/1445 | 1167/1441
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1441) | Canagliflozin 100 mg (N=1445) | Canagliflozin 300 mg (N=1441)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 7
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Pernicious Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 8 | 3 | 3
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 10 | 10 | 8
Adams-Stokes Syndrome (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 24 | 15 | 30
Angina Unstable (Cardiac disorders) | 20 | 24 | 28
Anginal Equivalent (Cardiac disorders) | 1 | 0 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1 | 1
Aortic Valve Stenosis (Cardiac disorders) | 1 | 1 | 1
Arrhythmia (Cardiac disorders) | 3 | 0 | 4
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 26 | 22 | 17
Atrial Flutter (Cardiac disorders) | 6 | 6 | 8
Atrioventricular Block (Cardiac disorders) | 2 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 2 | 2 | 3
Atrioventricular Block Second Degree (Cardiac disorders) | 3 | 2 | 2
Bradycardia (Cardiac disorders) | 4 | 2 | 5
Cardiac Arrest (Cardiac disorders) | 6 | 7 | 6
Cardiac Disorder (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure (Cardiac disorders) | 19 | 19 | 23
Cardiac Failure Acute (Cardiac disorders) | 2 | 1 | 0
Cardiac Failure Chronic (Cardiac disorders) | 5 | 3 | 2
Cardiac Failure Congestive (Cardiac disorders) | 20 | 15 | 14
Cardio-Respiratory Arrest (Cardiac disorders) | 2 | 3 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 2 | 4
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Cardiovascular Disorder (Cardiac disorders) | 1 | 1 | 1
Cor Pulmonale (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 24 | 24 | 23
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 2 | 2 | 0
Coronary Artery Stenosis (Cardiac disorders) | 5 | 5 | 7
Coronary Artery Thrombosis (Cardiac disorders) | 0 | 1 | 0
Hypertensive Heart Disease (Cardiac disorders) | 0 | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 2 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 2 | 1 | 2
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0 | 1
Myocardial Fibrosis (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 16 | 18 | 11
Myocardial Ischaemia (Cardiac disorders) | 9 | 11 | 6
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis Constrictive (Cardiac disorders) | 0 | 0 | 1
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0 | 0
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 0 | 2 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 2 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 6 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 2 | 1 | 1
Ventricular Fibrillation (Cardiac disorders) | 3 | 2 | 1
Ventricular Tachycardia (Cardiac disorders) | 3 | 2 | 3
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Developmental Hip Dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 2 | 4
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 3
Vertigo Positional (Ear and labyrinth disorders) | 2 | 1 | 1
Empty Sella Syndrome (Endocrine disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1
Hyperparathyroidism Primary (Endocrine disorders) | 0 | 1 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Amaurosis Fugax (Eye disorders) | 0 | 0 | 1
Blindness Unilateral (Eye disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 8 | 8 | 10
Cataract Diabetic (Eye disorders) | 0 | 0 | 1
Cataract Nuclear (Eye disorders) | 0 | 1 | 0
Cataract Subcapsular (Eye disorders) | 2 | 0 | 0
Dacryostenosis Acquired (Eye disorders) | 0 | 1 | 0
Diabetic Retinopathy (Eye disorders) | 1 | 3 | 2
Diplopia (Eye disorders) | 1 | 0 | 0
Exophthalmos (Eye disorders) | 1 | 0 | 0
Eye Haemorrhage (Eye disorders) | 1 | 1 | 1
Eyelid Ptosis (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 2 | 0 | 3
Lens Dislocation (Eye disorders) | 0 | 0 | 1
Macular Degeneration (Eye disorders) | 0 | 1 | 1
Macular Fibrosis (Eye disorders) | 1 | 0 | 1
Macular Hole (Eye disorders) | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 1 | 0
Ocular Myasthenia (Eye disorders) | 0 | 1 | 0
Open Angle Glaucoma (Eye disorders) | 0 | 0 | 1
Optic Ischaemic Neuropathy (Eye disorders) | 1 | 0 | 0
Retinal Detachment (Eye disorders) | 2 | 0 | 0
Retinal Vascular Thrombosis (Eye disorders) | 0 | 0 | 1
Retinopathy Proliferative (Eye disorders) | 0 | 1 | 1
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 1 | 0
Vitreous Floaters (Eye disorders) | 0 | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 2 | 1
Abdominal Hernia (Gastrointestinal disorders) | 3 | 2 | 5
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 3
Bowel Movement Irregularity (Gastrointestinal disorders) | 0 | 0 | 1
Chronic Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 2 | 0
Colitis Microscopic (Gastrointestinal disorders) | 1 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 2 | 0
Colon Dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1
Dieulafoy's Vascular Malformation (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 4 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Erosive Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 1
Gallstone Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Mucosal Hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 2
Gastrointestinal Erosion (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 4
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 2
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 3 | 0
Hernial Eventration (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 3 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 3 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Polyp (Gastrointestinal disorders) | 1 | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 2 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Achalasia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic Cyst (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic Pseudocyst (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 3 | 2
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 4 | 1
Pancreatitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 4 | 6 | 3
Rectal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 3
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 3 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 3 | 1
Varices Oesophageal (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Adverse Drug Reaction (General disorders) | 0 | 2 | 0
Application Site Dermatitis (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 2 | 0
Chest Discomfort (General disorders) | 3 | 3 | 2
Chest Pain (General disorders) | 23 | 26 | 13
Complication Associated with Device (General disorders) | 0 | 0 | 2
Death (General disorders) | 8 | 8 | 8
Drug Intolerance (General disorders) | 0 | 1 | 0
Facial Pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Generalised Oedema (General disorders) | 1 | 1 | 0
Impaired Healing (General disorders) | 0 | 2 | 0
Ischaemic Ulcer (General disorders) | 1 | 0 | 0
Medical Device Site Reaction (General disorders) | 0 | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 2
Necrosis (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 8 | 5
Oedema Peripheral (General disorders) | 3 | 3 | 1
Perforated Ulcer (General disorders) | 1 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 3
Strangulated Hernia (General disorders) | 0 | 0 | 1
Sudden Cardiac Death (General disorders) | 5 | 0 | 9
Sudden Death (General disorders) | 6 | 5 | 3
Vascular Stent Occlusion (General disorders) | 0 | 0 | 1
Vascular Stent Restenosis (General disorders) | 2 | 3 | 1
Alcoholic Liver Disease (Hepatobiliary disorders) | 1 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 2 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 5 | 5
Cholecystitis Acute (Hepatobiliary disorders) | 4 | 6 | 3
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 11 | 9 | 7
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder Disorder (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder Pain (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder Perforation (Hepatobiliary disorders) | 0 | 2 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0 | 2
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Fibrosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 0
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 1
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Portal Hypertension (Hepatobiliary disorders) | 0 | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 2 | 0 | 2
Post Cholecystectomy Syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Atopy (Immune system disorders) | 0 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Food Allergy (Immune system disorders) | 1 | 0 | 0
Abdominal Abscess (Infections and infestations) | 1 | 1 | 0
Abdominal Sepsis (Infections and infestations) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Abscess Limb (Infections and infestations) | 4 | 5 | 2
Anal Abscess (Infections and infestations) | 1 | 2 | 0
Appendicitis (Infections and infestations) | 2 | 3 | 6
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0
Arthritis Infective (Infections and infestations) | 1 | 2 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0 | 0
Biliary Sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 5 | 3
Bronchitis Bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0 | 0
Burn Infection (Infections and infestations) | 0 | 1 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Carbuncle (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 19 | 15 | 15
Cellulitis Gangrenous (Infections and infestations) | 0 | 1 | 2
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 3
Chronic Hepatitis B (Infections and infestations) | 0 | 1 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0
Colon Gangrene (Infections and infestations) | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1 | 1
Device Related Infection (Infections and infestations) | 1 | 1 | 2
Diabetic Foot Infection (Infections and infestations) | 1 | 2 | 6
Diabetic Gangrene (Infections and infestations) | 1 | 2 | 1
Diverticulitis (Infections and infestations) | 3 | 3 | 5
Endocarditis (Infections and infestations) | 0 | 0 | 1
Enterococcal Bacteraemia (Infections and infestations) | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 2
Erysipelas (Infections and infestations) | 1 | 3 | 5
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Eye Infection (Infections and infestations) | 1 | 1 | 0
Eye Infection Fungal (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 4 | 15 | 6
Gastroenteritis (Infections and infestations) | 6 | 5 | 8
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 2
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 1
Groin Abscess (Infections and infestations) | 1 | 0 | 0
Groin Infection (Infections and infestations) | 0 | 0 | 1
Haematoma Infection (Infections and infestations) | 1 | 1 | 0
Helicobacter Infection (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 2 | 1
Hiv Infection (Infections and infestations) | 1 | 0 | 0
Infected Cyst (Infections and infestations) | 0 | 1 | 1
Infected Dermal Cyst (Infections and infestations) | 0 | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 2 | 2 | 3
Infective Exacerbation of Bronchiectasis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 3 | 2
Intervertebral Discitis (Infections and infestations) | 0 | 1 | 1
Klebsiella Infection (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1 | 0
Localised Infection (Infections and infestations) | 1 | 4 | 10
Lower Respiratory Tract Infection (Infections and infestations) | 7 | 1 | 4
Lung Infection (Infections and infestations) | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 1 | 0
Medical Device Site Infection (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1
Meningitis Viral (Infections and infestations) | 0 | 1 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0 | 1
Nosocomial Infection (Infections and infestations) | 0 | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 7 | 11 | 12
Osteomyelitis Chronic (Infections and infestations) | 0 | 0 | 2
Otitis Externa (Infections and infestations) | 1 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pathogen Resistance (Infections and infestations) | 1 | 0 | 0
Pelvic Abscess (Infections and infestations) | 0 | 1 | 0
Penile Infection (Infections and infestations) | 0 | 1 | 0
Perineal Abscess (Infections and infestations) | 0 | 0 | 1
Perinephric Abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1 | 1
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Plasmodium Vivax Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 36 | 31 | 26
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia Influenzal (Infections and infestations) | 1 | 0 | 0
Post Procedural Cellulitis (Infections and infestations) | 0 | 0 | 1
Post Procedural Infection (Infections and infestations) | 1 | 2 | 3
Postoperative Abscess (Infections and infestations) | 0 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 5 | 2 | 4
Pseudomonal Bacteraemia (Infections and infestations) | 0 | 1 | 0
Psoas Abscess (Infections and infestations) | 0 | 1 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 3 | 3 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 0 | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0 | 0
Renal Tuberculosis (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 10 | 12 | 4
Septic Shock (Infections and infestations) | 3 | 0 | 2
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 2 | 1
Staphylococcal Abscess (Infections and infestations) | 0 | 0 | 2
Staphylococcal Infection (Infections and infestations) | 0 | 2 | 1
Staphylococcal Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 2 | 2
Streptococcal Bacteraemia (Infections and infestations) | 2 | 0 | 0
Streptococcal Infection (Infections and infestations) | 0 | 1 | 0
Streptococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 1
Superinfection Bacterial (Infections and infestations) | 0 | 0 | 1
Testicular Abscess (Infections and infestations) | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Typhoid Fever (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 16 | 15 | 6
Urosepsis (Infections and infestations) | 4 | 7 | 3
Vestibular Neuronitis (Infections and infestations) | 0 | 1 | 0
Viral Infection (Infections and infestations) | 1 | 3 | 2
Viral Pharyngitis (Infections and infestations) | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Vulval Abscess (Infections and infestations) | 1 | 0 | 0
Wound Abscess (Infections and infestations) | 0 | 1 | 0
Wound Infection (Infections and infestations) | 2 | 0 | 3
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 3 | 0 | 0
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 6 | 5
Arterial Bypass Occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arterial Bypass Stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1 | 3
Dural Tear (Injury, poisoning and procedural complications) | 0 | 1 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 4 | 4
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 7
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Foreign Body (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foreign Body in Eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture Displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 1 | 1
Heat Stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 3 | 4 | 7
Humerus Fracture (Injury, poisoning and procedural complications) | 2 | 4 | 8
Joint Dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 1 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Concussion Syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 2
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 3 | 8
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 | 1 | 2
Skin Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Skull Fractured Base (Injury, poisoning and procedural complications) | 0 | 1 | 2
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Spinal Cord Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Stomal Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 2
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 4 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular Graft Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 2 | 2
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 1 | 0
Blood Glucose Abnormal (Investigations) | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 1 | 1
Blood Pressure Abnormal (Investigations) | 0 | 0 | 1
Blood Pressure Decreased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1
Cardiac Stress Test Abnormal (Investigations) | 0 | 1 | 0
Catheterisation Cardiac (Investigations) | 0 | 1 | 0
Clostridium Test Positive (Investigations) | 0 | 1 | 0
Colonoscopy (Investigations) | 1 | 0 | 1
Electrocardiogram Abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram St Segment Depression (Investigations) | 0 | 0 | 1
Electrocardiogram St-T Segment Abnormal (Investigations) | 1 | 0 | 0
Exercise Test Abnormal (Investigations) | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 2 | 0
Precancerous Cells Present (Investigations) | 0 | 0 | 1
Renal Function Test Abnormal (Investigations) | 0 | 0 | 1
Troponin Increased (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 3 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 10 | 6 | 6
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 7 | 3 | 3
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 4 | 3
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hyperosmolar Hyperglycaemic State (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 12 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Ketosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 | 1 | 2
Metabolic Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 3 | 5 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Acquired Claw Toe (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4
Bone Atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diabetic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Gouty Tophus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 8 | 3
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 27 | 30 | 23
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Senile Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Appendix Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Benign Neoplasm of Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign Neoplasm of Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign Peritoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 0
Bladder Cancer Stage 0, with Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 6
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bronchial Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carcinoid Tumour of the Duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid Body Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chondrosarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 3
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Colon Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Head and Neck Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Kidney Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large Intestine Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 4
Lung Squamous Cell Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Small Intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Carcinoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Carcinoma of the Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Small Cell Lung Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Papillary Serous Endometrial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3
Penile Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 | 6
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Rectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Renal Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sarcoma Uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Squamous Cell Carcinoma of the Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Testicular Seminoma (Pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Transitional Cell Cancer of the Renal Pelvis and Ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Vulvovaginal Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Alcoholic Seizure (Nervous system disorders) | 0 | 0 | 1
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1
Basal Ganglia Infarction (Nervous system disorders) | 1 | 0 | 0
Basilar Artery Occlusion (Nervous system disorders) | 0 | 0 | 1
Brain Injury (Nervous system disorders) | 0 | 0 | 1
Brain Stem Haemorrhage (Nervous system disorders) | 1 | 0 | 0
Brain Stem Infarction (Nervous system disorders) | 0 | 0 | 2
Carotid Arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 5 | 5 | 11
Carotid Sinus Syndrome (Nervous system disorders) | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 2 | 2 | 2
Cerebellar Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebellar Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral Arteriosclerosis (Nervous system disorders) | 2 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 1 | 1
Cerebral Infarction (Nervous system disorders) | 3 | 2 | 2
Cerebrovascular Accident (Nervous system disorders) | 10 | 13 | 13
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 1 | 0
Cubital Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0 | 0
Diabetic Coma (Nervous system disorders) | 0 | 0 | 1
Diabetic Hyperosmolar Coma (Nervous system disorders) | 1 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 2 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Facial Paralysis (Nervous system disorders) | 0 | 0 | 1
Facial Paresis (Nervous system disorders) | 1 | 0 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 2 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0 | 0
Hyponatraemic Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Intercostal Neuralgia (Nervous system disorders) | 0 | 0 | 1
Intracranial Haematoma (Nervous system disorders) | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 4 | 3 | 2
Lacunar Infarction (Nervous system disorders) | 0 | 1 | 1
Lacunar Stroke (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 2 | 1 | 2
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Lumbosacral Radiculopathy (Nervous system disorders) | 0 | 1 | 1
Mental Impairment (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Motor Dysfunction (Nervous system disorders) | 0 | 0 | 1
Myasthenia Gravis (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 2 | 1
Orthostatic Intolerance (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Paralysis Recurrent Laryngeal Nerve (Nervous system disorders) | 0 | 1 | 0
Parkinson's Disease (Nervous system disorders) | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Partial Seizures (Nervous system disorders) | 0 | 1 | 0
Petit Mal Epilepsy (Nervous system disorders) | 0 | 0 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 2 | 3
Radiculopathy (Nervous system disorders) | 0 | 1 | 2
Reversible Cerebral Vasoconstriction Syndrome (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 2 | 2 | 1
Serotonin Syndrome (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spinal Claudication (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 7 | 9 | 5
Transient Ischaemic Attack (Nervous system disorders) | 15 | 7 | 16
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Vertebrobasilar Insufficiency (Nervous system disorders) | 3 | 2 | 1
Vertigo CNS Origin (Nervous system disorders) | 0 | 0 | 1
Vith Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1 | 0
Device Breakage (Product Issues) | 0 | 1 | 1
Device Damage (Product Issues) | 0 | 1 | 0
Affective Disorder (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Delirium Tremens (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2
Hallucination (Psychiatric disorders) | 1 | 1 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Major Depression (Psychiatric disorders) | 1 | 1 | 1
Mental Disorder (Psychiatric disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 4 | 2 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 1
Schizoaffective Disorder (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 1
Vascular Cognitive Impairment (Psychiatric disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 13 | 15 | 8
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder Prolapse (Renal and urinary disorders) | 0 | 0 | 2
Bladder Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Calculus Bladder (Renal and urinary disorders) | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 0 | 2
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 2 | 4
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 7 | 2 | 2
Oliguria (Renal and urinary disorders) | 1 | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 2 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 6 | 3
Renal Papillary Necrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 1 | 0 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Terminal Dribbling (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 1
Urethral Meatus Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1 | 4
Urinary Bladder Polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0 | 3
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 1
Acquired Phimosis (Reproductive system and breast disorders) | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 8 | 15
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 2
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Epididymal Cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Genital Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Orchitis Noninfective (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Pelvic Prolapse (Reproductive system and breast disorders) | 0 | 0 | 2
Prostatic Calcification (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 2 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 2
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0 | 2
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Uterovaginal Prolapse (Reproductive system and breast disorders) | 2 | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diaphragmatic Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 7
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 9
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Pulmonary Vein Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 4 | 9 | 10
Diabetic Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Guttate Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Keloid Scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Necrobiosis Lipoidica Diabeticorum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 | 10 | 14
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Arrhythmia Prophylaxis (Surgical and medical procedures) | 1 | 0 | 0
Fracture Treatment (Surgical and medical procedures) | 0 | 0 | 1
Gastric Bypass (Surgical and medical procedures) | 1 | 0 | 0
Hip Arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Incisional Hernia Repair (Surgical and medical procedures) | 1 | 0 | 0
Accelerated Hypertension (Vascular disorders) | 2 | 0 | 2
Aortic Aneurysm (Vascular disorders) | 4 | 2 | 0
Aortic Stenosis (Vascular disorders) | 1 | 3 | 3
Arterial Disorder (Vascular disorders) | 0 | 0 | 1
Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0
Arterial Thrombosis (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 2 | 1
Blood Pressure Inadequately Controlled (Vascular disorders) | 1 | 0 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 4 | 5
Dry Gangrene (Vascular disorders) | 1 | 0 | 2
Extremity Necrosis (Vascular disorders) | 0 | 1 | 4
Haematoma (Vascular disorders) | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 10 | 3 | 2
Hypertensive Crisis (Vascular disorders) | 4 | 5 | 3
Hypertensive Emergency (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 3 | 5 | 3
Iliac Artery Occlusion (Vascular disorders) | 0 | 1 | 0
Intermittent Claudication (Vascular disorders) | 3 | 3 | 4
Ischaemia (Vascular disorders) | 1 | 0 | 0
Leriche Syndrome (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Malignant Hypertension (Vascular disorders) | 1 | 0 | 1
Neurogenic Shock (Vascular disorders) | 0 | 2 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 4 | 12 | 11
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0 | 1
Peripheral Artery Occlusion (Vascular disorders) | 1 | 7 | 1
Peripheral Artery Stenosis (Vascular disorders) | 4 | 5 | 7
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 9 | 9 | 6
Peripheral Vascular Disorder (Vascular disorders) | 7 | 8 | 10
Subclavian Artery Stenosis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1 | 0
Varicose Vein (Vascular disorders) | 3 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1441) | Canagliflozin 100 mg (N=1445) | Canagliflozin 300 mg (N=1441)
Anaemia (Blood and lymphatic system disorders) | 55 | 41 | 40
Angina Pectoris (Cardiac disorders) | 36 | 25 | 30
Atrial Fibrillation (Cardiac disorders) | 38 | 38 | 29
Vertigo (Ear and labyrinth disorders) | 42 | 50 | 54
Cataract (Eye disorders) | 77 | 91 | 84
Diabetic Retinopathy (Eye disorders) | 46 | 45 | 50
Abdominal Pain (Gastrointestinal disorders) | 40 | 42 | 47
Abdominal Pain Upper (Gastrointestinal disorders) | 35 | 33 | 31
Constipation (Gastrointestinal disorders) | 61 | 73 | 70
Diarrhoea (Gastrointestinal disorders) | 119 | 105 | 147
Dyspepsia (Gastrointestinal disorders) | 46 | 43 | 32
Gastritis (Gastrointestinal disorders) | 31 | 44 | 38
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 32 | 41 | 46
Nausea (Gastrointestinal disorders) | 57 | 60 | 58
Toothache (Gastrointestinal disorders) | 31 | 38 | 32
Vomiting (Gastrointestinal disorders) | 39 | 42 | 39
Asthenia (General disorders) | 24 | 30 | 38
Chest Pain (General disorders) | 57 | 63 | 61
Fatigue (General disorders) | 57 | 59 | 59
Oedema Peripheral (General disorders) | 86 | 54 | 62
Pyrexia (General disorders) | 47 | 39 | 35
Thirst (General disorders) | 1 | 19 | 29
Hepatic Steatosis (Hepatobiliary disorders) | 32 | 18 | 20
Bronchitis (Infections and infestations) | 123 | 109 | 112
Cellulitis (Infections and infestations) | 26 | 37 | 37
Conjunctivitis (Infections and infestations) | 22 | 34 | 24
Cystitis (Infections and infestations) | 23 | 35 | 34
Gastroenteritis (Infections and infestations) | 42 | 54 | 43
Genital Infection Fungal (Infections and infestations) | 6 | 19 | 30
Influenza (Infections and infestations) | 86 | 100 | 82
Localised Infection (Infections and infestations) | 26 | 18 | 30
Lower Respiratory Tract Infection (Infections and infestations) | 33 | 32 | 28
Nasopharyngitis (Infections and infestations) | 220 | 225 | 203
Pharyngitis (Infections and infestations) | 31 | 43 | 24
Pneumonia (Infections and infestations) | 39 | 23 | 39
Sinusitis (Infections and infestations) | 45 | 58 | 65
Upper Respiratory Tract Infection (Infections and infestations) | 163 | 157 | 133
Urinary Tract Infection (Infections and infestations) | 128 | 132 | 159
Viral Infection (Infections and infestations) | 26 | 32 | 33
Vulvovaginal Mycotic Infection (Infections and infestations) | 10 | 30 | 31
Contusion (Injury, poisoning and procedural complications) | 34 | 38 | 36
Ligament Sprain (Injury, poisoning and procedural complications) | 24 | 33 | 19
Limb Injury (Injury, poisoning and procedural complications) | 33 | 31 | 26
Blood Creatine Phosphokinase Increased (Investigations) | 31 | 20 | 19
Blood Creatinine Increased (Investigations) | 28 | 33 | 35
Blood Pressure Increased (Investigations) | 35 | 17 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 91 | 55 | 63
Hypoglycaemia (Metabolism and nutrition disorders) | 174 | 181 | 210
Arthralgia (Musculoskeletal and connective tissue disorders) | 125 | 133 | 129
Back Pain (Musculoskeletal and connective tissue disorders) | 137 | 138 | 149
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 52 | 40 | 52
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 65 | 69 | 64
Myalgia (Musculoskeletal and connective tissue disorders) | 43 | 49 | 36
Neck Pain (Musculoskeletal and connective tissue disorders) | 22 | 20 | 30
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 84 | 83 | 83
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 98 | 105 | 92
Diabetic Neuropathy (Nervous system disorders) | 40 | 34 | 41
Dizziness (Nervous system disorders) | 33 | 34 | 61
Headache (Nervous system disorders) | 108 | 90 | 100
Hypoaesthesia (Nervous system disorders) | 19 | 34 | 24
Neuropathy Peripheral (Nervous system disorders) | 26 | 33 | 24
Depression (Psychiatric disorders) | 33 | 39 | 38
Insomnia (Psychiatric disorders) | 37 | 29 | 39
Dysuria (Renal and urinary disorders) | 15 | 30 | 32
Pollakiuria (Renal and urinary disorders) | 19 | 66 | 86
Balanoposthitis (Reproductive system and breast disorders) | 25 | 87 | 100
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 29 | 37 | 36
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 7 | 29 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 104 | 103 | 97
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 39 | 42
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 33 | 41 | 34
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 19 | 30
Rash (Skin and subcutaneous tissue disorders) | 28 | 38 | 45
Skin Lesion (Skin and subcutaneous tissue disorders) | 8 | 16 | 30
Skin Ulcer (Skin and subcutaneous tissue disorders) | 31 | 45 | 51
Hypertension (Vascular disorders) | 123 | 77 | 75
Hypotension (Vascular disorders) | 15 | 39 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT01032629/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT01032629/SAP_001.pdf